CLINICAL TRIAL: NCT00140426
Title: A Double-blind, Placebo Controlled Trial of Risperidone for the Treatment of Anorexia Nervosa
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Janssen Pharmaceuticals (Industry); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 03-0673; 5M01RR000069-45 (NIH)
Record Dates: First submitted 2005-08-31; First posted 2005-09-01 (Estimated); Results first posted 2016-02-02 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2015-12

CONDITIONS: Anorexia Nervosa
Keywords: Anorexia Nervosa; Risperidone; Atypical Neuroleptics; Dopamine; Leptin; Body Image; Adolescents
MeSH Terms: conditions — Anorexia Nervosa | interventions — Risperidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator): double blind study of risperidone for anorexia nervosa. this is the subject group that receives placebo.
  Interventions: Drug: Placebo
- risperidone (Active Comparator): Study is double blind, placebo controlled. This is the subject group on active medication
  Interventions: Drug: Risperidone

INTERVENTIONS:
Drug: Risperidone — risperidone titrated 0.5 to 4 mg over study enrollment. Mean Length of Phase 1 is currently 10 weeks.
  Other Names: Risperdal
  Arms: risperidone
Drug: Placebo — Comparison of risperidone versus placebo for the treatment of symptoms related to anorexia nervosa.
  Other Names: placebo - inactive pill
  Arms: placebo

SUMMARY:
The aim of this pilot study is to determine the safety and efficacy of risperidone for the treatment of anorexia nervosa.

Hypothesis 1: Subjects on risperidone will show a more significant decrease in body image distortion and Eating Disorder Inventory -2 scores than subjects on placebo.

Hypothesis 2: Subjects on risperidone will reach and maintain at or above 90% Ideal body weight sooner than controls.

DETAILED DESCRIPTION:
The lack of effective medications for the symptoms of anorexia nervosa (AN), combined with early promising findings in case reports (Risperidone and Olanzapine) and one open study of olanzapine have led to increased use of these medications for individuals with AN. This double-blind placebo controlled study of risperidone will attempt to determine if risperidone is effective in decreasing core symptoms of anorexia nervosa and decreasing the length of time required to reach and maintain at or about 90% Ideal body weight. The safety of risperidone in this population will also be examined through monitoring of Extrapyramidal Symptoms, Tardive Dyskinesia, Electrocardiograms's, Resting Energy Expenditure, liver enzymes and other blood chemistry. Other possible variables which may mediate the recovery process or be impacted by risperidone,such as leptin and anxiety symptoms are also being measured.

ELIGIBILITY:
Inclusion Criteria:

* Primary Diagnosis of Anorexia Nervosa
* Female, age 12-21
* Active in a level of care for AN at The Children's Hospital, Denver
* As long as there is a primary dx of AN, co-morbid diagnoses may be included.
* If taking an antidepressant, must be on a stable dose for 3 weeks prior to entering the study, and dose of antidepressant may not be changed during Phase 1 of the study.
* If choosing to discontinue antidepressant medication, must be off the medication for 3 weeks prior to beginning the study.
* If sexually active, must use birth control during the study and have a monthly pregnancy test.

Exclusion Criteria:

* Previous enrollment in this study on a prior admission
* Previous allergic reaction to risperidone or other atypical neuroleptic
* Positive pregnancy test
* Neurologic disorder other than benign essential tremor
* Taking a psychotropic medication other than antidepressant and discontinuing the medication is not recommended.
* Active hepatic or renal disease
* Wards of the state
* Males

Ages: 12 Years to 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2004-08; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer O Hagman, MD, Principal Investigator — University of Colorado, Health Sciences Center and The Children's Hospital, Denver
Locations (1):
- The Children's Hospital, Denver, Colorado, United States

REFERENCES:
- [Derived] Hagman J, Gralla J, Sigel E, Ellert S, Dodge M, Gardner R, O'Lonergan T, Frank G, Wamboldt MZ. A double-blind, placebo-controlled study of risperidone for the treatment of adolescents and young adults with anorexia nervosa: a pilot study. J Am Acad Child Adolesc Psychiatry. 2011 Sep;50(9):915-24. doi: 10.1016/j.jaac.2011.06.009. Epub 2011 Aug 5. PMID 21871373

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: double blind study of risperidone for anorexia nervosa. this is the subject group that receives placebo.
  Risperidone or placebo: risperidone titrated 0.5 to 4 mg over study enrollment. Mean Length of Phase 1 is currently 10 weeks.
- Risperidone: Study is double blind, placebo controlled. This is the subject group on active medication
  Risperidone: Comparison of risperidone versus placebo for the treatment of symptoms related to anorexia nervosa. Titration of study medication from 0.5 to 4 mg based on weight gain to target IBW.
Period: Overall Study
Arm/Group | Placebo | Risperidone
Started | 22 | 19
Completed | 22 | 16
Not Completed | 0 | 3
Not completed — Withdrawal by Subject | 0 | 3

BASELINE CHARACTERISTICS:
Population: Females age 12 - 21
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Risperidone | Total
Number analyzed (Participants) | 22 | 19 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 19 | 13 | 32
  Between 18 and 65 years | 3 | 6 | 9
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.8 (2.3) | 16.2 (2.5) | 15.98 (2.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 19 | 41
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 22 | 19 | 41

OUTCOME MEASURES:

1. Primary Outcome: Change in Eating Disorder Inventory-2 Drive for Thinness Subscale (DT)
Description: Eating Disorder Inventory -2 - Subscale : Drive for Thinness Subscale (DT). Lower scores are better on this scale and indicate less cognitive focus on drive for thinness.
  The EDI 2 is a 91 item scale with 8 subscales - (Drive for thinness, Bulimia, body dissatisfaction, ineffectiveness, perfection, interpersonal distrust, interoceptive awareness and maturity fears.). The DT subscale was used for this outcome. Respondents rate each item as "usually , often, sometimes, rarely or never". Subscale scores are computed by summing all item scores for each subscale. There are 7 items in the DT subscale (questions 1,7,11,16,25,32 and 49). the subscale score range is 0-21. The EDI-2 was completed by subjects at baseline and then monthly during study participation (range 0 -18 weeks). Change in the DT subscale score was calculated using an estimate of change in score between week 0 and week 7 derived from the mixed effect model across all time points.
Time Frame: month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Risperidone
Number analyzed (Participants) | 22 | 16
units on a scale | 1.36 (5.09) | 3.93 (6.95)

2. Primary Outcome: Change in Eating Disorder Inventory (EDI)-2 Score for Body Dissatisfaction (BD)
Description: change in Eating Disorder Inventory (EDI) 2-score for Body Dissatisfaction (BD).
  Lower scores are better on this scale. Higher scores indicate the subject has greater body dissatisfaction. BD is one of the 8 subscales of the EDI-2. 9 of the 91 questions in the EDI-2 scale constitute this subscale. The score range is 0-27. Subjects completed the EDI-2 at baseline and monthly during study participation (range 0 to 18 weeks). Change in the BD subscale score during the study was calculated using an estimate of change in score between week 0 and week 7 derived from the mixed effect model across all time points.
Time Frame: monthly
Population: 1 risperidone subject was missing data for BD at this data point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Risperidone
Number analyzed (Participants) | 22 | 15
units on a scale | 0.82 (5.96) | 2.67 (7.93)

3. Primary Outcome: Hazard Ratio for Time to Reaching Ease Of Eating Level 3 From Start of Study (Normal Eating Behavior)
Description: The Ease of Eating Scale (EOES) is a 14 item scale which measures Food avoidance behaviors (FABs). The scale is rated by staff observing a subject eating a meal or snack. 0 = normal eating behavior, maximum score 28.
  Higher scores indicate more food avoidance behaviors, such as taking small bites, taking > 30 seconds between bites (slow eating), etc.
  EOE was completed for each meal a subject ate in the program and scores were averaged for each week in the study and entered in the data base.
  Change in EOES score was calculated by evaluating change over time. This measure was only used in Phase 1 of the study, for days the subjects were in the treatment program.
Time Frame: weekly up to study endpoint: reaching target weight and maintaining for 1 month
Population: 2 patients in the placebo group were treated as inpatients and had no EOE data.
Measure: Number (95% Confidence Interval); unit: hazard ratio
Groups:
- Risperidone: Study is double blind, placebo controlled. This is the subject group on active medication.
  Risperidone: Comparison of risperidone versus placebo for the treatment of symptoms related to anorexia nervosa. Titration of study medication from 0.5 to 4 mg based on weight gain to target IBW.
Arm/Group | Placebo | Risperidone
Number analyzed (Participants) | 20 | 16
hazard ratio | 0.85 [0.41 to 1.74] | 1 [1 to 1]
Statistical Analysis 1: Comparison: Placebo vs Risperidone; Test type: Superiority or Other; p = 0.55, Regression, Cox; Time to reaching ease of eating level 3 assessed using Cox regression as some patients did not reach it during the study; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.41 to 1.74] — The hazard ratio is for the placebo group versus the treatment group. A hazard ratio <1 implies that the placebo group had a lower risk of achieving EOE level 3, although not statistically significant. Achieving EOE level 3 was the desired endpoint

4. Secondary Outcome: Time to Reach 90% Ideal Body Weight (IBW) and Maintain for 1 Month, Stratified by >=80% at Start of Study
Description: The mean survival time and its standard error were underestimated because the largest observation was censored and the estimation was restricted to the largest event time. These estimates were produced using Kaplan-Meier probabilities. This was measured weekly from 0-18 weeks.
Time Frame: weekly
Measure: Mean (Standard Error); unit: weeks
Arm/Group | Placebo | Risperidone
Number analyzed (Participants) | 10 | 6
weeks | 10.7 (1.6) | 8.1 (0.2)

5. Secondary Outcome: Change in Ratings of Anxiety Symptoms on the Multidimensional Anxiety Scale for Children (MASC)
Description: The Multidimensional Anxiety Scale for Children (MASC) is a self report measure completed by the subject that measures anxiety symptoms.
  Higher scores indicate greater anxiety. A score of over 50 is significant for anxiety
  Change in MASC scores was calculated using an estimate of change in score between week 0 and week 7 derived from the mixed effect model across all time points.
Time Frame: monthly to study end point
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Risperidone
Number analyzed (Participants) | 18 | 15
units on a scale | 7.41 (7.87) | 7.87 (11.19)

6. Secondary Outcome: Change in Leptin Levels
Description: Leptin levels were measured by serum blood draws, results reports in nanograms / ml (ng/ml).
Time Frame: Week 0 and week 7
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Placebo | Risperidone
Number analyzed (Participants) | 19 | 12
ng/ml | 0.88 (4.13) | 3.27 (3.04)

7. Secondary Outcome: Change in Prolactin Levels
Description: Prolactin serum blood levels, measured in nanograms / ml
Time Frame: week 0 and week 7
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Placebo | Risperidone
Number analyzed (Participants) | 19 | 12
ng/ml | -5.18 (5.89) | 38.27 (33.05)
Statistical Analysis 1: Comparison: Placebo vs Risperidone; Test type: Superiority or Other; p = 0.10, t-test, 2 sided; Mean Difference (Net) = -2.38, Standard Deviation 3.74
Statistical Analysis 2: Comparison: Placebo vs Risperidone; Test type: Superiority or Other; p < 0.01, t-test, 2 sided; Mean Difference (Final Values) = -43.45, Standard Deviation 20.88

8. Secondary Outcome: Time to Reach 90% IBW and Maintain for 1 Month, Stratified by IBW <80% at Start of Study
Description: The mean survival time and its standard error were underestimated because the largest observation was censored and the estimation was restricted to the largest event time. These estimates were produced using Kaplan-Meier probabilities.
Time Frame: 0 - 18 weeks
Measure: Mean (Standard Error); unit: weeks
Groups:
- Placebo: double blind study of risperidone for anorexia nervosa. this is the subject group that receives placebo.
  This subject group received placebo tablets which appeared identical to risperidone
- Risperidone: Study is double blind, placebo controlled. This is the subject group on active medication
  Risperidone: this group of patients received the active study medication. Titration of study medication from 0.5 to 4 mg based on weight gain to target IBW.
Arm/Group | Placebo | Risperidone
Number analyzed (Participants) | 12 | 12
weeks | 10.1 (0.4) | 12.9 (1.3)

9. Primary Outcome: Color A Person Test (CAPT)
Description: Color A Person Test (CAPT) - Subjects color an outlined image of a body to indicate body dissatisfaction (red (5)= very dissatisfied, Yellow, dissatisfied, black, neutral, green satisfied, blue very satisfied (1). The outline is divided into16 sections for scoring. The CAPT was completed at baseline and monthly during study participation.
  Total CAPT scores were calculated by adding the total score and dividing by 16. Score range is 1-5. Lower scores indicate less body dissatisfaction.
  Change in the CAPT score during the study was calculated using an estimate of change in score between week 0 and week 7 derived from the mixed effect model across all time points.
Time Frame: monthly
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Risperidone or Placebo: double blind study of risperidone for anorexia nervosa. this is the subject group that receives placebo.
  Risperidone or placebo: risperidone titrated 0.5 to 4 mg over study enrollment. Mean Length of Phase 1 is currently 10 weeks.
Arm/Group | Risperidone or Placebo | Risperidone
Number analyzed (Participants) | 22 | 18
units on a scale | 0.03 (0.75) | 0.22 (0.79)
Statistical Analysis 1: Comparison: Risperidone or Placebo vs Risperidone; Null hypothesis: no difference in change from baseline to end of treatment for CAPT total score; Test type: Superiority or Other; p = 0.47, t-test, 2 sided; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-0.71 to 0.33], Standard Error of Mean 0.26 — The mean difference was for placebo - risperidone

10. Primary Outcome: Body Image Software (BIS): Average Distortion
Description: Body Image Software (BIS) - the subject adjusts a digital image of themselves on the computer using the direction to "adjust their image to how they see themselves right now", this determines their perception of their current image. Accuracy is measured by a smaller score between desired image and actual image.
  Change in the BIS Average Distortion score during the study was calculated using an estimate of change in score between week 0 and week 7 derived from the mixed effect model across all time points.
  There are no identifiable minimum/maximum values as there would be in a questionnaire scale. There are no subscales. The BIS program calculates the difference between their actual image and the size of the image they have adjusted the digital image to based on their perception of "how they see themselves right now"
Time Frame: monthly
Population: Change from baseline to end of study was compared between arms. Some patients did not complete this outcome measurement.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Risperidone or Placebo | Risperidone
Number analyzed (Participants) | 21 | 16
units on a scale | -0.22 (8.75) | 1.40 (8.36)
Statistical Analysis 1: Comparison: Risperidone or Placebo vs Risperidone; Test type: Superiority or Other; p = 0.57, t-test, 2 sided

11. Primary Outcome: Body Image Software (BIS): Average Desired Thinness
Description: Body Image Software (BIS) - the subject adjusts a digital image of themselves on the computer to "their desired image". The BIS program calculates the difference between their actual image, and how much they have adjusted the image to represent their "desired image". Accuracy is measured by a smaller score between desired image and actual image.
  Change in BIS - Average Desired Thinness score was calculated using an estimate of change in score between week 0 and week 7 derived from the mixed effect model across all time points.
  There are no identifiable minimum/maximum values as there would be in a questionnaire scale. . There are no subscales.
Time Frame: monthly
Population: Many patients did not complete this outcome measurement. Change from baseline to end of study were compared between arms.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Risperidone or Placebo | Risperidone
Number analyzed (Participants) | 10 | 7
units on a scale | 1.88 (9.24) | -1.42 (10.31)
Statistical Analysis 1: Comparison: Risperidone or Placebo vs Risperidone; Test type: Superiority or Other; p = 0.50, t-test, 2 sided

12. Primary Outcome: Body Image Software (BIS) - Point of Subjective Equality (PSE)
Description: Body Image Software (BIS) - the subject adjusts a digital image of themselves on the computer to their desired image, and also completes a task that determines their perception of their current image. Accuracy is measured by a smaller score between desired image and actual image.
  Change in BIS -PSE was calculated using an estimate of change in score between week 0 and week 7 derived from the mixed effect model across all time points.
  There are no identifiable minimum/maximum values as there would be in a questionnaire scale. Interpreting the PSE is how it compares to a PSE = 0, which is no distortion in body size.
Time Frame: monthly
Population: Change from baseline to end of study was compared between arms. Some patients did not complete this outcome measurement.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Risperidone or Placebo | Risperidone
Number analyzed (Participants) | 19 | 16
units on a scale | -0.32 (5.81) | -2.18 (7.92)
Statistical Analysis 1: Comparison: Risperidone or Placebo vs Risperidone; Test type: Superiority or Other; p = 0.43, t-test, 2 sided

13. Primary Outcome: Body Image Software (BIS) - Difference Limen (DL)
Description: Body Image Software (BIS) - the subject adjusts a digital image of themselves on the computer to their desired image, and also completes a task that determines their perception of their current image. Accuracy is measured by a smaller score between desired image and actual image.
  Change in BIS-DL was calculated using an estimate of change in score between week 0 and week 7 derived from the mixed effect model across all time points.
  There are no identifiable minimum/maximum values as there would be in a questionnaire scale. There are no subscales. Interpreting the DL occurs by referencing it to DL= 0, which would reflect a total inability to detect size differences, which has never occurred in studies using the BIS program.
Time Frame: monthly
Population: Change from baseline to end of study was compared between arms. Some patients did not complete this outcome measurement.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Risperidone or Placebo | Risperidone
Number analyzed (Participants) | 19 | 16
units on a scale | -0.19 (1.10) | -1.16 (2.18)
Statistical Analysis 1: Comparison: Risperidone or Placebo vs Risperidone; Test type: Superiority or Other; p = 0.12, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: While patients were on the study medication (placebo or risperidone)
Arm/Group | Placebo | Risperidone
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/18
Other Adverse Events (participants affected / at risk) | 17/22 | 16/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=22) | Risperidone (N=18)
Fatigue (Nervous system disorders) | 8 (22) | 11 (39)
dizziness (Nervous system disorders) | 4 (4) | 4 (15)
gastrointestinal complaints (Gastrointestinal disorders) | 13 (53) | 7 (35)
headache (Nervous system disorders) | 8 (8) | 4 (5)
Depression (Psychiatric disorders) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 3 (6) | 1 (1)
insomnia (Nervous system disorders) | 2 (4) | 0 (0)
Extrapyramidal symptoms (EPS) (Musculoskeletal and connective tissue disorders) | 8 (46) | 8 (19) — Measured on the Simpson rating scale
Tardive dyskinesia (Nervous system disorders) | 1 (2) | 6 (14) — as measured by the Abnormal Involuntary Movement Scale (AIMS)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes